CLINICAL TRIAL: NCT00703131
Title: A Single-center Single Arm Prospective Study Evaluating the Surgisis Biodesign Anal Fistula Plug
Brief Title: Surgisis Anal Fistula Plug Study: An Experience in Saudi Arabia
Acronym: SurgiSIS AFP
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-012
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Anal Fistula
Keywords: fistula; anal fistula
MeSH Terms: conditions — Rectal Fistula; Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Anal Fistula Plug
  Interventions: Device: Anal Fistula Plug (SurgiSIS AFP)

INTERVENTIONS:
Device: Anal Fistula Plug (SurgiSIS AFP) — Anal Fistula Plug
  Other Names: SurgiSIS Biodesign

SUMMARY:
The Surgisis Anal Fistula Plug study is a clinical trial conducted in Saudi Arabia to study the safety and effectiveness of the Surgisis AFP Plug in the treatment of chronic anal fistulas.

DETAILED DESCRIPTION:
Up to 30 patients will be treated with the Surgisis Anal Fistula Plug using a standardized surgical procedure to plug their anal fistula. Patients will be followed periodically until their 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Primary, persistent, or recurrent fistula tract that is either transsphincteric, suprasphincteric, or extrasphincteric
* Signed informed consent
* Willing to return for follow-up visits

Exclusion Criteria:

* Crohn's Disease
* Ulcerative Colitis
* HIV Positive
* Immune System Disorder
* Collagen Disorder
* Tuberculosis
* History of radiation to anorectal region
* Allergies to pig tissue
* Religious or cultural objection to use of pig tissue in this surgical application
* J-pouch fistulas
* Previous Surgisis AFP Plug placement in target fistula tract
* Tracts with acute abscess, infection or inflammation
* Superficial fistula tracts conventionally treated with fistulotomy/fistulectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Saudi Arabia with chronic anal fistula
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Healing Success | 12 months

SECONDARY OUTCOMES:
Change in Quality of Life Measures | 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Zubaidi, MD, Principal Investigator — King Khalid University Hospital
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia